CLINICAL TRIAL: NCT00810407
Title: Special Investigation For Non-hiv Patients Of Mycobutin (Regulatory Post Marketing Commitment Plan).
Brief Title: Safety And Efficacy Of Rifabutin In Patients For Non-HIV Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0061006
Record Dates: First submitted 2008-12-09; First posted 2008-12-18 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-11

CONDITIONS: Tuberculosis; Non-tuberculous Mycobacterial Diseases (Including MAC Disease)
MeSH Terms: conditions — Tuberculosis | interventions — Rifabutin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rifabutin: Patients administered Rifabutin.
  Interventions: Drug: rifabutin

INTERVENTIONS:
Drug: rifabutin — Mycobutin® capsules150mg depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. " 1.Tuberculosis : The usual adult dosage for oral use is 150 mg to 300 mg of rifabutin once daily.For the treatment of multiple-drug resistance tuberculosis, the usual dosage for oral use is 300 to 450 mg of rifabutin once daily.
  2.Treatment of non-tuberculous mycobacterial diseases (including MAC disease) : The usual adult dosage for oral use is 300 mg of rifabutin once daily".
  Other Names: Mycobutin.

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Mycobutin® should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Mycobutin® in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Mycobutin®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A0061006 prescribes the Mycobutin®).
Sampling Method: Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0061006&StudyName=Safety%20And%20Efficacy%20Of%20Rifabutin%20In%20Patients%20For%20Non-HIV%20Patients%0A

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 628 subjects were registered in this study. Of the 628 subjects, 594 subjects CRFs were collected and included in the study. Of the 594 subjects, 6 subjects were excluded from the safety analysis set (SAS). In total, 588 subjects were included in the SAS as the completed the study
Groups:
- Mycobutin (Rifabutin): Participants who received Mycobutin as indicated in the approved local product document were observed for a period of 1 year. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Mycobutin (Rifabutin)
Started | 594
Completed | 588
Not Completed | 6
Not completed — Protocol Violation | 3
Not completed — No Visit After First Day of Treatment | 3

BASELINE CHARACTERISTICS:
Population: A total of 588 participants received Mycobutin at least once in this study. Of the 594 participants, 6 participants were excluded from the baseline analysis due to following reasons: protocol violation and no visit after first day of treatment.
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 588
Age, Customized [Count of Participants; unit: Participants]
  <15 years | 1
  ≥15 and <65 years | 234
  ≥65 years | 349
  Unknown | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 363
  Male | 225
Diagnosis [Count of Participants; unit: Participants]
  Tuberculosis | 134
  Mycobacterium Avium Complex (MAC) | 428
  Non-tuberculous Mycobacteria Other Than MAC | 19
  Coinfection | 5
  Others | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Mycobutin in a participant who received Mycobutin. Relatedness to Mycobutin was assessed by the physician/investigator.
Time Frame: 1 year
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received Mycobutin at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 588
Participants
  Treatment-Related Adverse Event | 387
  Treatment-Related Serious Adverse Event | 113

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Mycobutin in a participant who received Mycobutin. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to Mycobutin was assessed by the physician/investigator.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 588
Participants | 71

3. Primary Outcome: Number of Participants With Treatment-Related Adverse Events by Diagnosis
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Mycobutin in a participant who received Mycobutin. Relatedness to Mycobutin was assessed by the physician/investigator. Participants with treatment related adverse events were counted by diagnosis to assess whether they were risk factors for the treatment related adverse events.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 588
Participants
  Tuberculosis: number analyzed (Participants) | 134
  Tuberculosis | 60
  Mycobacterium Avium Complex (MAC): number analyzed (Participants) | 428
  Mycobacterium Avium Complex (MAC) | 312
  Non-tuberculous Mycobacteria Other Than MAC: number analyzed (Participants) | 19
  Non-tuberculous Mycobacteria Other Than MAC | 11
  Coinfection: number analyzed (Participants) | 5
  Coinfection | 4
  Others: number analyzed (Participants) | 2
  Others | 0
Statistical Analysis 1: Comparison: Mycobutin (Rifabutin); The factor tested was "diagnosis". The null hypothesis was that there was no association between diagnosis and the number of participants with treatment-related adverse events; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Primary Outcome: Number of Participants With Treatment-Related Adverse Events by Gender
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Mycobutin in a participant who received Mycobutin. Relatedness to Mycobutin was assessed by the physician/investigator. Participants with treatment related adverse events were counted by gender to assess whether they were risk factors for the treatment related adverse events.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 588
Participants
  Female: number analyzed (Participants) | 363
  Female | 264
  Male: number analyzed (Participants) | 225
  Male | 123
Statistical Analysis 1: Comparison: Mycobutin (Rifabutin); The factor tested was "gender". The null hypothesis was that there was no association between gender and the number of participants with treatment-related adverse events; Test type: Superiority or Other; p < 0.001, Fisher Exact

5. Primary Outcome: Number of Participants With Treatment-Related Adverse Events by Age
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Mycobutin in a participant who received Mycobutin. Relatedness to Mycobutin was assessed by the physician/investigator. Participants with treatment related adverse events were counted by age to assess whether they were risk factors for the treatment related adverse events.
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 588
Participants
  <15 years: number analyzed (Participants) | 1
  <15 years | 1
  ≥15 and <65 years: number analyzed (Participants) | 234
  ≥15 and <65 years | 149
  ≥65 years: number analyzed (Participants) | 349
  ≥65 years | 235
  Unknown: number analyzed (Participants) | 4
  Unknown | 2
Statistical Analysis 1: Comparison: Mycobutin (Rifabutin); The factor tested was "age". The null hypothesis was that there was no association between age of participants and the number of participants with treatment-related adverse events; Test type: Superiority or Other; p = 0.587, Fisher Exact
Statistical Analysis 2: Comparison: Mycobutin (Rifabutin); The factor tested was "age". The null hypothesis was that there was no ordinal trend in the number of participants with treatment-related adverse events across the age at baseline; Test type: Superiority or Other; p = 0.428, Cochran-Armitage (EXACT)

6. Primary Outcome: Clinical Efficacy Rate
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Clinical effectiveness of Mycobutin was assessed as "effective," "ineffective," or "unassessable" by the physician/investigator. Overall effectiveness of Mycobutin was determined by the physician/investigator based on clinical symptoms, laboratory values, and other examinations such as bacterial values.
Time Frame: 1 year
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician/investigator based upon change in clinical symptoms and laboratory findings) at least once.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 332
Percentage of Participants | 62.7 [57.2 to 67.9]

7. Primary Outcome: Clinical Efficacy Rate by Diagnosis
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Clinical effectiveness of Mycobutin was assessed as "effective," "ineffective," or "unassessable" by the physician/investigator. Overall effectiveness of Mycobutin was determined by the physician/investigator based on clinical symptoms, laboratory values, and other examinations such as bacterial values. Participants achieved clinical effectiveness by diagnosis were counted to assess whether they contribute to the clinical effectiveness.
Time Frame: 1 year
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician/investigator based upon change in clinical symptoms and laboratory findings) at least once. Participants with observed effectiveness data were included in table.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 332
Percentage of Participants
  Tuberculosis: number analyzed (Participants) | 96
  Tuberculosis | 82.3 [73.2 to 89.3]
  Mycobacterium Avium Complex (MAC): number analyzed (Participants) | 219
  Mycobacterium Avium Complex (MAC) | 53.9 [47.0 to 60.6]
  Non-tuberculous Mycobacteria Other Than MAC: number analyzed (Participants) | 12
  Non-tuberculous Mycobacteria Other Than MAC | 58.3 [27.7 to 84.8]
  Coinfection: number analyzed (Participants) | 4
  Coinfection | 100.0 [39.8 to 100.0]
  Others: number analyzed (Participants) | 1
  Others | 0.0 [0.0 to 97.5]

8. Primary Outcome: Clinical Efficacy Rate by Gender
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of Mycobutin was assessed as "effective," "ineffective," or "unassessable" by the physician/investigator. Overall effectiveness of Mycobutin was determined by the physician/investigator based on clinical symptoms, laboratory values, and other examinations such as bacterial values. Participants achieved clinical effectiveness by gender were counted to assess whether they contribute to the clinical effectiveness.
Time Frame: 1 year
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 332
Percentage of Participants
  Male: number analyzed (Participants) | 149
  Male | 71.1
  Female: number analyzed (Participants) | 183
  Female | 55.7

9. Primary Outcome: Clinical Efficacy Rate by Age
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of Mycobutin was assessed as "effective," "ineffective," or "unassessable" by the physician/investigator. Overall effectiveness of Mycobutin was determined by the physician/investigator based on clinical symptoms, laboratory values, and other examinations such as bacterial values. Participants achieved clinical effectiveness by age were counted to assess whether they contribute to the clinical effectiveness.
Time Frame: 1 year
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Mycobutin (Rifabutin)
Number analyzed (Participants) | 332
Percentage of Participants
  ˂15 years: number analyzed (Participants) | 1
  ˂15 years | 0.0
  ≥15 and <65 years: number analyzed (Participants) | 131
  ≥15 and <65 years | 71.8
  ≥65 years: number analyzed (Participants) | 196
  ≥65 years | 57.1
  Unknown: number analyzed (Participants) | 4
  Unknown | 50

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Mycobutin (Rifabutin)
Serious Adverse Events (participants affected / at risk) | 184/588
Other Adverse Events (participants affected / at risk) | 470/588
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mycobutin (Rifabutin) (N=588)
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 12
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 12
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 10
Liver disorder (Hepatobiliary disorders) | 20
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Chills (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 18
Oedema peripheral (General disorders) | 1
Platelet count decreased (Investigations) | 10
Neutrophil count decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 11
Aspergillus infection (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Mycobacterium avium complex infection (Infections and infestations) | 4
Osteomyelitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 3
Pneumonia pseudomonal (Infections and infestations) | 1
Pulmonary mycosis (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 5
Bone marrow failure (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Tonic convulsion (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Optic neuropathy (Eye disorders) | 1
Uveitis (Eye disorders) | 12
Visual acuity reduced (Eye disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Cardiac failure acute (Cardiac disorders) | 2
Cardiogenic shock (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1
Gastrointestinal amyloidosis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3
Abortion (Pregnancy, puerperium and perinatal conditions) | 1
Death (General disorders) | 2
Drug interaction (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mycobutin (Rifabutin) (N=588)
Liver disorder (Hepatobiliary disorders) | 29
Pyrexia (General disorders) | 62
Anaemia (Blood and lymphatic system disorders) | 19
Leukopenia (Blood and lymphatic system disorders) | 18
Decreased appetite (Metabolism and nutrition disorders) | 52
Diarrhoea (Gastrointestinal disorders) | 23
Nausea (Gastrointestinal disorders) | 18
Hepatic function abnormal (Hepatobiliary disorders) | 66
Drug eruption (Skin and subcutaneous tissue disorders) | 21
Rash (Skin and subcutaneous tissue disorders) | 27
Gamma-glutamyltransferase increased (Investigations) | 19
Platelet count decreased (Investigations) | 54
White blood cell count decreased (Investigations) | 62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.